CLINICAL TRIAL: NCT01146288
Title: Effect of Acetazolamide and Furosemide on Obesity-induced Glomerular Hyperfiltration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, boris zingerman, MD, Rabin Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ObesAceta 1
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2015-06-04 (Estimated); Status verified 2015-06

CONDITIONS: Obesity-induced Hyperfiltration
Keywords: obesity; acetazolamide; furosemide
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Furosemide first, then Acetazolamide (Experimental): Two renal function studies will be performed: one before and after intravenous furosemide and the second before and after intravenous acetazolamide. Participants will receive intravenous furosemide 2 mg/5min or intravenous acetazolamide 5 mg/kg/5 min.
  Interventions: Drug: Furosemide first, then Acetazolamide
- Acetazolamide first, then Furosemide (Experimental): Two renal function studies will be performed: one before and after intravenous acetazolamide and the second before and after intravenous furosemide. Participants will receive intravenous furosemide 2 mg/5min or intravenous acetazolamide 5 mg/kg/5 min.
  Interventions: Drug: Acetazolamide first, then Furosemide

INTERVENTIONS:
Drug: Furosemide first, then Acetazolamide — Two renal function studies will be performed: one before and after intravenous furosemide and the second before and after intravenous acetazolamide. Subjects will receive 300 mg of lithium carbonate at 22.00 the day before the renal function tests. A priming dose of inulin (50 mg/kg) and p-aminohippuric acid (8 mg/kg) will be administered and a 200-300 ml p.o water load will be given. Thereafter, inulin and p-aminohippuric acid will be infused continuously. After the first 60 minutes, 8 accurately timed urine collections of 30 to 40 minutes will be obtained by spontaneous voiding. After the first 4 timed urine collections, participants will receive intravenous furosemide 2 mg/5min or intravenous acetazolamide 5 mg/kg/5 min.Four other times urine collections will be performed thereafter.
  Arms: Furosemide first, then Acetazolamide
Drug: Acetazolamide first, then Furosemide — Two renal function studies will be performed: one before and after intravenous acetazolamide and the second before and after intravenous furosemide. Subjects will receive 300 mg of lithium carbonate at 22.00 the day before the renal function tests.A priming dose of inulin (50 mg/kg) and p-aminohippuric acid (8 mg/kg) will be administered and a 200-300 ml p.o water load will be given. Thereafter, inulin and p-aminohippuric acid will be infused continuously. After the first 60 minutes, 8 accurately timed urine collections of 30 to 40 minutes will be obtained by spontaneous voiding. After the first 4 timed urine collections, participants will receive intravenous furosemide 2 mg/5min or intravenous acetazolamide 5 mg/kg/5 min.Four other times urine collections will be performed thereafter.
  Arms: Acetazolamide first, then Furosemide

SUMMARY:
Background:

Obesity is associated with a high prevalence of chronic kidney disease.The glomerular hyperfiltration associated with obesity may play a role in the pathogenesis of obesity associated chronic kidney disease. Attenuation of hyperfiltration by pharmacological means may slow down the development and progression of chronic renal failure. The investigators have previously shown that acetazolamide, a proximally acting diuretic that activates tubuloglomerular feedback(TGF) by increasing solute delivery to the Macula DENSA, abates glomerular hyperfiltration. The present study was designed to test the hypothesis that this decrease in hyperfiltration is specific to acetazolamide and not due to a non specific diuretic effect. The aim of the present study is to compare the effects of furosemide and acetazolamide on glomerular hemodynamics in subjects with severe obesity.

Methods:

A randomized double-blind crossover controlled design will be used. Fifteen obese subjects and ten subjects with normal body weight will participate in the study. Obese subjects will undergo measurement of glomerular filtration rate (GFR)(inulin clearance), renal plasma flow (RPF) (p-aminohippuric acid clearance), filtration fraction, fractional excretion of lithium (FE LI) and blood pressure, before and after intravenous administration of furosemide 2 mg. and acetazolamide 5 mg/kg BW. Ten subjects with normal body weight will undergo measurement of renal function without administration of diuretics.

DETAILED DESCRIPTION:
BACKGROUND Almost half of the causes of death in the industrial world are due to cardio-vascular (CV) disease. Two of the main risk factors for CV disease have become much more prevalent during the last decades, reaching epidemic dimensions in the 21st century: hypertension and obesity. In 2003-2004, 66% of the adult USA population had a body mass index(BMI)over 25, while 32% had a BMI over 30 .Hypertension is more prevalent in obese than in lean subjects .The cause and effect relationship between these two conditions is supported by the fact that weight loss is associated with a decrease in blood pressure .

Salt retention by the kidney is one of the important mechanisms involved in the pathogenesis of hypertension in obesity. Studies in animal models and in humans showed that increased salt reabsorption occurs in the tubules in obesity. Another renal functional abnormality occurring in obesity is glomerular hyperfiltration, characterized by increased renal plasma flow (RPF) and increased glomerular filtration rate(GFR) up to twice the normal level . The structural basis to these functional abnormalities is renal hypertrophy and glomerular enlargement.

These functional and structural abnormalities have deleterious consequences:

1. Increased urinary albumin excretion. Microalbuminuria, an important risk factor for CV disease, has a high prevalence in obese subjects .
2. Increased risk for the development of focal segmental glomerulosclerosis, the so-called obesity related glomerulopathy. The incidence of this disease has multiplied 10 times within 15 yrs in the USA .
3. Increased rate of progression of chronic renal insufficiency in kidney disease not primarily caused by obesity. Following initial glomerular damage from any cause, the number of remnant functioning glomeruli decreases. The consequent compensatory increase in single nephron filtration rate of these remnant glomeruli leads to further glomerular damage in kidney disease not related to obesity . In the obese with chronic renal damage, the obesity related hyperfiltration amplifies the compensatory augmentation in single nephron GFR of remnant nephrons, thus worsening glomerular damage, irrespective of the cause of the primary insult.

The clinical relevance of these abnormalities is reflected in the sharp increase in the risk of developing end stage renal disease in the obese. This relative risk, independently of confounders as diabetes mellitus, hypertension and dyslipidemia, is 3 to 5 depending on the severity of obesity .

Considering the role of hyperfiltration in the pathogenesis of chronic kidney disease (CKD) in the obese, attenuation of hyperfiltration by pharmacological means may slow down the development and progression of chronic renal failure. One of the tools available is activating tubuloglomerular feedback (TGF). Tubuloglomerular feedback (TGF) refers to the alterations in GFR that can be induced by changes in tubular flow rate. An increase in the delivery of chloride to the Macula DENSA results in a reduction in GFR, resulting in a decrease in the tubular flow rate delivered to the Macula DENSA. An increase in chloride delivery to the Macula DENSA can be obtained by administrating acetazolamide, a diuretic acting on the proximal tubule. We have previously shown that administration of acetazolamide to obese subjects results in attenuation of glomerular hyperfiltration.

The aim of the present study is to show that the effect of acetazolamide on GFR is specific and not due to its diuretic effect. We will study the effects of furosemide, a diuretic which does not activate TGF ,on GFR and RPF in obese subjects in comparison with acetazolamide.

Methods:

A 24-hour urine collection will be performed during the week prior to the renal function test studies for assessment of sodium intake.

Obese subjects: A randomized double-blind crossover controlled design will be used. Two renal function studies will be performed: one before and after intravenous furosemide and the second before and after intravenous acetazolamide. Subjects will receive 300 mg of lithium carbonate at 22.00 the day before the renal function tests. They will be instructed to drink 250 ml of water at bedtime. Renal function tests will start at 08.00 a.m. after a 10-hour fast, excepting a drink of 250 ml of water at 07.00 a.m. Intravenous catheters will be placed in each upper limb for infusion of clearance markers and blood sampling. After blood sampling for urea, creatinine, proteins, glucose, electrolytes, blood gases, insulin, renin, aldosterone, Hba1c, CBC. A priming dose of inulin (50 mg/kg) and p-aminohippuric acid (8 mg/kg) will be administered and a 200-300 ml p.o water load will be given. Thereafter, inulin and p-aminohippuric acid will be infused continuously. After the first 60 minutes, 8 accurately timed urine collections of 30 to 40 minutes will be obtained by spontaneous voiding. Peripheral venous blood will be drawn to bracket each urine collection. Arterial pressure will be measured by a trained observer, after 30 minutes of rest in the supine position, using an electronic oscillometric blood pressure measuring device. The cuff will be appropriately sized to the diameter of the arm and the arm positioned at the heart level. At least 8 measurements will be performed during the study, each measurement being the mean of 3 readings. After the first 4 timed urine collections, participants will receive intravenous furosemide 2 mg/5min or intravenous acetazolamide 5 mg/kg/5 min. Four other times urine collections will be performed thereafter. Subjects will be randomized to receive during the first study either furosemide or acetazolamide. The second study will be performed one to two weeks after the first study, using the drug that had not administrated during the first study.

Subjects with normal body weight: will undergo measurement of renal function without administration of diuretics (one renal function study, same protocol like obese subjects, with 4 urine collections only).

Laboratory procedures: Plasma and urinary concentrations of inulin and p-aminohippuric acid will be analyzed by colorimetric methods .Lithium in serum and urine will be measured . Urine microalbumin will be determined by competitive chemiluminescent enzyme immunoassay .

Calculations: GFR will be determined from the average value for the timed inulin clearances, and renal plasma flow (RPF) - from the average value for the timed p-aminohippurate clearances. The fractional excretion of lithium (FE Li) will be calculated as lithium clearance / GFR, using two timed urine collections. FE Li will be determined as the average value for these two measurements Statistical Analysis: The significance of differences between groups will be evaluated by paired and unpaired two-tailed Student's t-test. The Student's t-test will be applied to non-normally distributed data (albumin excretion rate and fractional lithium excretion) after log transformation. P<0.05 will be considered as significant. The response to treatment with furosemide will be compared to the response to treatment with acetazolamide using ANOVA.

ELIGIBILITY:
Inclusion Criteria:

* 15 obese men (BMI>30), aged 18 to 55, with glomerular hyperfiltration (creatinine clearance>130 ml/min)) and 10 normal body weight men (BMI<25), aged 18 to 55.

Exclusion Criteria:

* Heart failure, CKD, COPD
* Known allergy to furosemide, acetazolamide, inulin or amino-hippurate
* Pharmacologic treatment for hypertension, cardiac disease, diabetes mellitus
* Treatment with corticosteroids, antiepileptics or NSAID

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-07; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris Zingerman, MD, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

REFERENCES:
- [Derived] Conley MM, McFarlane CM, Johnson DW, Kelly JT, Campbell KL, MacLaughlin HL. Interventions for weight loss in people with chronic kidney disease who are overweight or obese. Cochrane Database Syst Rev. 2021 Mar 30;3(3):CD013119. doi: 10.1002/14651858.CD013119.pub2. PMID 33782940
- [Derived] Zingerman B, Herman-Edelstein M, Erman A, Bar Sheshet Itach S, Ori Y, Rozen-Zvi B, Gafter U, Chagnac A. Effect of Acetazolamide on Obesity-Induced Glomerular Hyperfiltration: A Randomized Controlled Trial. PLoS One. 2015 Sep 14;10(9):e0137163. doi: 10.1371/journal.pone.0137163. eCollection 2015. PMID 26367377

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants recruited between July 2010 and October 2012.
Pre-assignment Details: 19 screened, 6 excluded (2 did not meet inclusion criteria, 2 refused participation, 2 unable to adequately collect urine).
Groups:
- Acetazolamide First, Then Furosemide: Intravenous acetazolamide 5 mg/kg/5 min. in first intervention period and intravenous furosemide 2 mg/5min in second intervention period (after washout period).
- Furosemide First , Than Acetazolamide: Intravenous furosemide 2 mg/5min in first intervention period and intravenous acetazolamide 5 mg/kg/5 min. in second intervention period (after washout period).
Period: First Intervention(1 Day)
Arm/Group | Acetazolamide First, Then Furosemide | Furosemide First , Than Acetazolamide
Started | 7 | 6
Completed | 7 | 5
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1
Period: Second Intervention (1 Day)
Arm/Group | Acetazolamide First, Then Furosemide | Furosemide First , Than Acetazolamide
Started | 7 | 5
Completed | 7 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Acetazolamide First, Then Furosemide: intravenous acetazolamide 5 mg/kg/5 min. in first intervention period, intravenous furosemide 2 mg/5min in second intervention period (after washout period).
- Furosemide First, Then Acetazolamide: intravenous furosemide 2 mg/5min. in first intervention period, intravenous acetazolamide 5 mg/kg/5 min. in second intervention period (after washout period).
- Total: Total of all reporting groups
Arm/Group | Acetazolamide First, Then Furosemide | Furosemide First, Then Acetazolamide | Total
Number analyzed (Participants) | 7 | 5 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 5 | 12
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Standard Deviation); unit: years] | 37 (6.6) | 36 (7.1) | 36 (8)
Sex/Gender, Customized [Number; unit: participants]
  male | 7 | 5 | 12

OUTCOME MEASURES:

1. Primary Outcome: Change in GFR (ml/Min)
Time Frame: baseline and after diuretics administration
Measure: Mean (Standard Deviation); unit: ml/min
Groups:
- Acetazolamide: intravenous acetazolamide 5 mg/kg/5 min.
- Furosemide: intravenous furosemide 2 mg/5min.
Arm/Group | Acetazolamide | Furosemide
Number analyzed (Participants) | 12 | 12
ml/min
  GFR before acetazolamide/furosemide administration | 151 (22) | 152 (18)
  GFR after acetazolamide/furosemide administration | 120 (16) | 150 (28)

2. Primary Outcome: Renal Vascular Resistance (mm Hg/[ml/Min])
Time Frame: baseline and after diuretics administration
Measure: Mean (Standard Deviation); unit: mm Hg/[ml/min]
Arm/Group | Acetazolamide | Furosemide
Number analyzed (Participants) | 12 | 12
mm Hg/[ml/min]
  before acetazolamide/furosemide administration | 0.078 (1.017) | 0.073 (0.010)
  after acetazolamide/furosemide administration | 0.088 (0.021) | 0.080 (0.019)

ADVERSE EVENTS:
Groups:
- P-aminohippuric Acid: Intravenous priming dose of p-aminohippuric acid (8 mg/kg) before diuretics administration
Arm/Group | Acetazolamide | Furosemide | P-aminohippuric Acid
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1/13
Other Adverse Events (participants affected / at risk) | 3/12 | 0/12 | 0/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide (N=0) | Furosemide (N=0) | P-aminohippuric Acid (N=13)
angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) — angioedema after p-aminohippuric acid administration, before diuretics administration
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acetazolamide (N=12) | Furosemide (N=12) | P-aminohippuric Acid (N=12)
hand paresthesia (General disorders) | 2 (2) | 0 (0) | 0 (0) — hand paresthesia following acetazolamide administration
lip parestesia (General disorders) | 1 (1) | 0 (0) | 0 (0) — lip paresthesia following acetazolamide administration
alteration of the sense of taste (General disorders) | 1 (1) | 0 (0) | 0 (0) — alteration of the sense of taste after acetazolamide administration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes